## Prevalence and characteristics of somatic symptom disorder in the elderly in a community-based population: a large-scale cross-sectional study in China

## Assessment of Somatic Symptom in Chinese Community-Dwelling People

| Protocol Number | SSSCN202011 |
|-----------------|--------------|
| NCT No. | NCT04815863 |
| Date | Sep 20, 2018 |

## STUDY PROTOCOL SYNOPSIS

| Title | Prevalence and characteristics of somatic symptom disorder in the |
|---|---|
| Title | , , |
| | elderly in a community-based population: a large-scale cross- |
| ~ | sectional study in China |
| Sponsor | Investigator-Initiated Trial (IIT) |
| Primary Objectives | 1. to clarify the prevalence of somatic symptom disorder (SSD), |
| | depressive disorders, and anxiety disorders in the elderly in China; |
| | 2. to identify physical and psychological differences between the |
| | elderly and non-elderly; |
| | 3. to explore risk factors for SSD in the elderly. |
| Study Design | This prospective cross-sectional study (Assessment of Somatic |
| | Symptom in Chinese Community-Dwelling People, |
| | ClinicalTrials.gov identifier NCT04815863, registered on |
| | 06/12/2020) is a multicenter registry conducted in Shanghai, China, |
| | under the supervision of the Shanghai Association of Chinese |
| | Integrative Medicine. |
| | A multistage and stratified systematic sampling technique will be |
| | used to choose representative districts from sixteen districts in |
| | Shanghai, which are then divided into low, medium, and high |
| | economic levels according to the per capita gross domestic product |
| | of each district in 2018. Eleven districts will be selected |
| | proportionally and randomly and represented by 105 community |
| | health service institutions. The study was approved by institutional |
| | review committees at each center. The study is compliant with the |
| | 1975 Declaration of Helsinki guidelines. |
| | (1) assessment of somatic symptom disorder (SSD) |
| | The Somatic Symptom questionnaire is self-administered with an |
| | abbreviated 20-item measure. Briefly, it is composed of four |
| | dimensions: physical disorders, depressive disorders, anxiety |
| | disorders and depressive and anxiety disorders. Half of the items ask |
| | about physical complaints (one item per body system). SSS-CN |
| | scores ranging from 20 to 29, 30–39, 40–59 and $\geq$ 60 correspond to |
| | normal, mild, moderate and severe SSD, respectively. |
| | (2) assessment of depressive and anxiety disorders |
| | All participants will be assessed for depressive and anxiety |
| | disorders according to the PHQ-9 and GAD-7, which evaluate the |
| | frequencies at which certain symptoms had been experienced over |
| | the last two weeks, ranging from 0 ('not at all') to 3 ('nearly every |
| | day'). The cutoff values are listed below. For PHQ-9, scores of 5–9 |
| | indicate mild depressive disorder, 10–14 indicate moderate |
| | depressive disorder, 15–19 indicate moderately severe depressive |
| | disorder and≥20 indicate severe depressive disorder. For GAD-7, |
| | scores range from 0 to 21, with scores of 5–9, $10$ – $14$ , and $\ge 15$ |

| | representing mild, moderate, and severe anxiety symptom levels, |
|---|---|
| | respectively. |
| | (3) sociodemographic and clinical characteristics |
| | Sociodemographic data, including age, gender, level of education |
| | and marital status, will also be collected. A semi-structured |
| | questionnaire concerning clinical characteristics will be administered |
| | to survey participants' medical and medication histories. |
| Number of | Enrollment: 9110 [anticipate] |
| Subjects | Elderly group: 6874 [anticipate] |
| | Non-elderly group: 2236 [anticipate] |
| Enrollment | Inclusion criteria were: |
| Criteria | (1) voluntary participation and provision of written consent to |
| | participate in the study's evaluation and assessment; |
| | (2) completion of the SSS-CN questionnaire, Patient Health |
| | Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder-7 |
| | (GAD- 7) questionnaires. |
| | Exclusion criteria were : |
| | (1) patients lacking self-assessed abilities or who refused to |
| | participate; |
| | (2) patients who have been previously confirmed to have serious |
| | mental disorders, mental retardation, or dementia; |
| | (3) patients with cancer or central nervous system diseases; |
| | (4) patients with any missing data within questionnaire items or with |
| | more than one item missing from sociodemographic information; |
| | (5) patients with any medical conditions that in the opinion of the |
| | investigators will not be appropriate to participate in the study. |
| Safety Assessment | Adverse events were not required in this study protocol. |
| <b>Endpoints</b> | Number of Participants With Somatic Symptoms Disorder |
| Liupoints | 2. Number of Participants With Somatic Symptoms Disorder |
| | Accompanied With Anxiety |
| | 3. Number of Participants With Somatic Symptoms Disorder |
| Statistical | Accompanied With Depression |
| Statistical | Descriptive statistics for each group, such as counts and percentages |
| Analysis | (%) for non-continuous variables, will be reported for all |
| | sociodemographic and clinical characteristics. The prevalences of |
| | SSD of various severities for different genders and for participants |
| | diagnosed with depressive and anxiety disorders will be calculated. |
| | In order to assess whether SSD, depressive and anxiety disorders are |
| | associated with aged groups and whether depressive and anxiety |
| | disorders are associated with the severity of SSD, binary logistic |
| | regressions will be performed, adjusting for gender, educational |
| | level (middle school and below, high school, college, master and |
| | above), marital status (never married, married, divorced, widowed), |
| | hypertension (yes/no), diabetes mellitus (yes/ no), CV disease |

(yes/no), endocrine and metabolic disease except DM (yes/no), other diseases (yes/no), surgery (yes/no) and antipsychotic intake (yes/no) in all models.

Univariate analyses and binary logistic regression models will be used to assess the effects of sociodemographic factors and clinical characteristics on SSD in the non- elderly and elderly. Categorical sociodemographic and clinical variables will be analyzed by chisquare test. Binary logistic regressions will be performed using SSD (yes/no) as the dependent variable, adjusting for gender, educational level, marital status, and antipsychotic intake.

Fisher's exact test was used instead of the chi-square test only when one or more expectations for each cell of the 2-by-2 tables was below 5. A significance level was set at a p-value < 0.05 (two-tailed). Missing data were imputed with a multiple imputation approach. All statistical analyses were performed with SPSS 22 (IBM SPSS Statistics for Windows, Version 22.0. Armonk, NY: IBM Corp).